CLINICAL TRIAL: NCT05777590
Title: Prospective Comparison of ICG Microangiography and Conventional Angiography in Severe Frostbite
Brief Title: Comparison of ICG Microangiography and Conventional Angiography in Severe Frostbite
Status: Active, not recruiting | Type: Observational
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Other Study IDs: A22-321
Record Dates: First submitted 2023-01-14; First posted 2023-03-21 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Frostbite
Keywords: Frostbite; Angiogram; Indocyanine Green; ICG
MeSH Terms: conditions — Frostbite

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Indocyanine Green Angiogram — Angiogram using ICG dye the occurs directly after conventional angiogram in assessment of frostbite patients undergoing thrombolysis
  Other Names: ICG

SUMMARY:
Severe frostbite injury is a significant cause of morbidity in northern climates. Minnesota has some of the highest numbers of severe frostbite injuries in North America. As a result, Regions Hospital has the best opportunity to study this disease process and improve outcomes for frostbite patients. The diagnostic methods for severe frostbite injury vary from institution to institution and there is no standard practice. Commonly utilized methods include conventional angiography, Technetium 99 triple phase bone scans, SPECT studies, Indocyanine Green microangiography, and doppler studies. The proposed pilot study aims to directly compare conventional angiography imaging to ICG microangiography in adult patients with severe frostbite. Severe frostbite is defined as 4th degree: frostbite resulting in vascular occlusion and tissue ischemia. Both imaging modalities have been used for the diagnosis and monitoring of severe frostbite injury but there has never been a study directly comparing these two imaging modalities.

DETAILED DESCRIPTION:
Frostbite injury has been a significant cause of morbidity and mortality for as long as humans have experienced cold winters. When frostbite occurs, there are two primary mechanisms through which tissue damage occurs, though the main mechanism focused on here is systemic cooling. Frostbite is a multiphase process that starts with systemic cooling. As the body cools, blood is shunted from the extremities to the core to maintain heat in the vital organs. During this shunting, there is extensive vasospasm in the extremities and the tissue becomes ischemic. Upon further cooling, tissue ice crystals form within the cells and interstitial spaces causing desiccation and cell destruction. This occurs in the soft tissues and also affects the endothelium of the micro- and macro-vasculature. Clots form in the microvasculature, worsening the ischemia. All ischemic tissues release pro-inflammatory factors, which increase inflammation and worsen clotting.

Upon rewarming of the frozen tissues, the reperfusion can worsen the inflammatory state as these factors released by the ischemic tissue are now able to circulate. Rapid rewarming is used as a tool to mitigate this reperfusion injury, but it does not eliminate the damage. After rapid rewarming, the tissue is assessed for the extent of damage to determine next treatment steps. Diagnosis varies by institution, but the main goal of all diagnostic modalities is to determine if there is a vascular cutoff causing tissue ischemia.

At Regions Hospital, the main diagnostic method that has been used for over 20 years is conventional angiography. This clearly demonstrates the microvasculature of the tissues and allows the intra-arterial catheter directed sheaths to be placed to start thrombolytics, heparin, and vasodilators to treat the tissue ischemia. Other diagnostic modalities used elsewhere include Technetium 99 triple phase bone scans, SPECT imaging, and indocyanine green (ICG) microangiography. All of these imaging modalities demonstrate the perfusion of the affected tissue but do not allow for directed delivery of thrombolytics. In institutions that use these imaging techniques, thrombolytics are typically delivered in an intravenous fashion rather than intra-arterial.

ICG microangiography is a technology that has had rapidly expanding applications in recent decades. These have included retinal imaging, determining perfusion of colorectal anastomoses, biliary imaging, and assessing the blood supply of tissue flaps. It has recently been used in diagnosis of frostbite with good correlation with severe final amputation levels. It is easy to use, non-radiating, can be performed at the bedside, and cheaper than other imaging modalities.

Given that every hospital has different diagnostic and treatment algorithms, these different imaging modalities have rarely been compared in the same patient. The current best metric is comparing the imaging modality with the amount of tissue that is amputated as demonstrated in prior studies cited here. This research application provides a unique opportunity to compare two imaging modalities head-to-head in the same patient and determine their concordance or discordance.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (>18 years old) patients
2. Diagnosed with severe frostbite by conventional angiography
3. Undergoing thrombolysis with catheter directed lytics
4. Clinically sober at the time of consent
5. Cognitively able to provide consent as determined by clinician's best judgement
6. Normal kidney function (GFR >60)

Exclusion Criteria:

1. Pregnant. Pregnancy will be determined by standard of care pregnancy test performed on all female frostbite patients who are receiving lytics.
2. Iodine allergy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing conventional angiography and thrombolysis for severe frostbite. will be identified by the burn surgeons and advance practice practitioners. They will evaluate the patients to determine whether they meet the inclusion/exclusion criteria of the study.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2023-02-03 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of Angiography and ICG microangiography imaging demonstrating ischemic tissue present in severe frostbite scored by Hennepin Frostbite Score. | Through study completion, an average of 2 years
  Hypothesize that these two imaging modalities (ICG (indocyanine green) and conventional angiography) will be concordant at demonstrating the ischemic tissue present in severe frostbite.

SECONDARY OUTCOMES:
Safety of indocyanine green when delivered in close association with contrast dye (used in conventional angiography) measured by number of adverse events | Through study completion, an average of 2 years
  Contrast dye used in conventional angiography is associated with nephrotoxicity and other risks. Indocyanine green dye is generally considered to be a highly safe product with minimal risks associated with administration. It has been used for decades with minimal side effects. It is hypothesized that ICG dye will not result in any increase in risk to the patient when delivered in temporal proximity to conventional dye.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Lacey, MD, Principal Investigator — Regions Hospital
Locations (1):
- Regions Hospital, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lacey AM, Rogers C, Endorf FW, Fey RM, Gayken JR, Schmitz KR, Punjabi GV, Whitley AB, Masters TC, Moore JC, Nygaard RM. An Institutional Protocol for the Treatment of Severe Frostbite Injury-A 6-Year Retrospective Analysis. J Burn Care Res. 2021 Aug 4;42(4):817-820. doi: 10.1093/jbcr/irab008. PMID 33484248
- [Background] Gonzaga T, Jenabzadeh K, Anderson CP, Mohr WJ, Endorf FW, Ahrenholz DH. Use of Intra-arterial Thrombolytic Therapy for Acute Treatment of Frostbite in 62 Patients with Review of Thrombolytic Therapy in Frostbite. J Burn Care Res. 2016 Jul-Aug;37(4):e323-34. doi: 10.1097/BCR.0000000000000245. PMID 25950290
- [Background] Gao Y, Wang F, Zhou W, Pan S. Research progress in the pathogenic mechanisms and imaging of severe frostbite. Eur J Radiol. 2021 Apr;137:109605. doi: 10.1016/j.ejrad.2021.109605. Epub 2021 Feb 17. PMID 33621855
- [Background] Millet JD, Brown RK, Levi B, Kraft CT, Jacobson JA, Gross MD, Wong KK. Frostbite: Spectrum of Imaging Findings and Guidelines for Management. Radiographics. 2016 Nov-Dec;36(7):2154-2169. doi: 10.1148/rg.2016160045. Epub 2016 Aug 5. PMID 27494386
- [Background] Twomey JA, Peltier GL, Zera RT. An open-label study to evaluate the safety and efficacy of tissue plasminogen activator in treatment of severe frostbite. J Trauma. 2005 Dec;59(6):1350-4; discussion 1354-5. doi: 10.1097/01.ta.0000195517.50778.2e. PMID 16394908
- [Background] Heard J, Shamrock A, Galet C, Pape KO, Laroia S, Wibbenmeyer L. Thrombolytic Use in Management of Frostbite Injuries: Eight Year Retrospective Review at a Single Institution. J Burn Care Res. 2020 May 2;41(3):722-726. doi: 10.1093/jbcr/iraa028. PMID 32030427
- [Background] Masters T, Omodt S, Gayken J, Logue C, Westgard B, Hendriksen S, Walter J, Nygaard R. Microangiography to Monitor Treatment Outcomes Following Severe Frostbite Injury to the Hands. J Burn Care Res. 2018 Jan 1;39(1):162-167. doi: 10.1097/BCR.0000000000000526. PMID 28328661
- [Background] Lacey AM, Fey RM, Gayken JR, Endorf FW, Schmitz KR, Punjabi GV, Masters TC, Nygaard RM. Microangiography: An Alternative Tool for Assessing Severe Frostbite Injury. J Burn Care Res. 2019 Aug 14;40(5):566-569. doi: 10.1093/jbcr/irz112. PMID 31298700
- [Background] WEATHERLEY-WHITE RC, SJOSTROM B, PATON BC. EXPERIMENTAL STUDIES IN COLD INJURY. II. THE PATHOGENESIS OF FROSTBITE. J Surg Res. 1964 Jan;4:17-22. doi: 10.1016/s0022-4804(64)80004-4. No abstract available. PMID 14106388
- [Background] Rohrer MJ, Natale AM. Effect of hypothermia on the coagulation cascade. Crit Care Med. 1992 Oct;20(10):1402-5. doi: 10.1097/00003246-199210000-00007. PMID 1395660
- [Background] Zook N, Hussmann J, Brown R, Russell R, Kucan J, Roth A, Suchy H. Microcirculatory studies of frostbite injury. Ann Plast Surg. 1998 Mar;40(3):246-53; discussion 254-5. doi: 10.1097/00000637-199803000-00009. PMID 9523607
- [Background] Bourne MH, Piepkorn MW, Clayton F, Leonard LG. Analysis of microvascular changes in frostbite injury. J Surg Res. 1986 Jan;40(1):26-35. doi: 10.1016/0022-4804(86)90141-1. PMID 3941548
- [Background] Robson MC, Heggers JP. Evaluation of hand frostbite blister fluid as a clue to pathogenesis. J Hand Surg Am. 1981 Jan;6(1):43-7. doi: 10.1016/s0363-5023(81)80010-x. PMID 7204918
- [Background] McCauley RL, Hing DN, Robson MC, Heggers JP. Frostbite injuries: a rational approach based on the pathophysiology. J Trauma. 1983 Feb;23(2):143-7. PMID 6827634
- [Background] Rogers C, Lacey AM, Endorf FW, Punjabi G, Whitley A, Gayken J, Fey R, Schmitz K, Nygaard RM. The Effects of Rapid Rewarming on Tissue Salvage in Severe Frostbite Injury. J Burn Care Res. 2022 Jul 1;43(4):906-911. doi: 10.1093/jbcr/irab218. PMID 34791315
- [Background] Braun JD, Trinidad-Hernandez M, Perry D, Armstrong DG, Mills JL Sr. Early quantitative evaluation of indocyanine green angiography in patients with critical limb ischemia. J Vasc Surg. 2013 May;57(5):1213-8. doi: 10.1016/j.jvs.2012.10.113. Epub 2013 Jan 24. PMID 23352361
- [Background] Jafari MD, Lee KH, Halabi WJ, Mills SD, Carmichael JC, Stamos MJ, Pigazzi A. The use of indocyanine green fluorescence to assess anastomotic perfusion during robotic assisted laparoscopic rectal surgery. Surg Endosc. 2013 Aug;27(8):3003-8. doi: 10.1007/s00464-013-2832-8. Epub 2013 Feb 13. PMID 23404152
- [Background] Zhi Z, Yin X, Dziennis S, Wietecha T, Hudkins KL, Alpers CE, Wang RK. Optical microangiography of retina and choroid and measurement of total retinal blood flow in mice. Biomed Opt Express. 2012 Nov 1;3(11):2976-86. doi: 10.1364/BOE.3.002976. Epub 2012 Oct 24. PMID 23162733
- [Background] Nygaard RM, Whitley AB, Fey RM, Wagner AL. The Hennepin Score: Quantification of Frostbite Management Efficacy. J Burn Care Res. 2016 Jul-Aug;37(4):e317-22. doi: 10.1097/BCR.0000000000000277. PMID 26536540

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT05777590/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-10): https://cdn.clinicaltrials.gov/large-docs/90/NCT05777590/ICF_001.pdf